CLINICAL TRIAL: NCT07340489
Title: Chemoradiotherapy Combined With Serplulimab for Locally Advanced Cervical Cancer: A Prospective, Multicenter, Randomized, Phase II Clinical Trial
Brief Title: Serplulimab for Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20251312
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; immunotherapy; chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: chemotherapy combined with immunotherapy and radiotherapy (Experimental): chemotherapy an Serplulimab plus chemoradiotherapy group
  Interventions: Drug: Serplulimab; Radiation: radiotherapy; Drug: Chemotherapy
- Control group: immunotherapy and radiotherapy (Placebo Comparator): Serplulimab plus chemoradiotherapy group
  Interventions: Drug: Serplulimab; Radiation: radiotherapy

INTERVENTIONS:
Drug: Serplulimab — intravenous infusion of 300 mg, administered every 3 weeks as one cycle, on the first day of each cycle, with a maximum treatment duration of 2 years (up to 35 treatment cycles)
Radiation: radiotherapy — Pelvic external beam radiotherapy was delivered with a prescribed dose of 45.0-50.4 Gy in 25-28 fractions to the PTV, administered once daily, five days per week; the PGTVnd received a simultaneous integrated boost to 53.50-59.92 Gy in 25-28 fractions. During radiotherapy, concurrent chemotherapy with weekly cisplatin was administered.
  Brachytherapy was delivered with 28 Gy in 4 fractions, prescribed to the 100% isodose line covering the CTV.
Drug: Chemotherapy — Two cycles of induction chemotherapy were administered prior to concurrent chemoradiotherapy, consisting of cisplatin 60-75 mg/m² on days 1 and 2 of each cycle, once every 3 weeks (21 days), and nab-paclitaxel 135-175 mg/m² by intravenous infusion on day 1 of each cycle, once every 3 weeks (21 days). After completion of concurrent chemoradiotherapy, patients received four cycles of consolidation chemotherapy using the same cisplatin and nab-paclitaxel regimen as above.
  Arms: Experimental: chemotherapy combined with immunotherapy and radiotherapy

SUMMARY:
This study is a randomized, controlled, open-label, phase II clinical trial designed to enroll patients with previously untreated locally advanced cervical cancer. The study aims to evaluate the efficacy and safety of adding chemotherapy to serplulimab combined with concurrent chemoradiotherapy. The primary endpoint of this study is progression-free survival (PFS).

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label, phase II clinical trial designed to evaluate the efficacy and safety of serplulimab in combination with chemotherapy and concurrent chemoradiotherapy in patients with locally advanced cervical cancer. Eligible patients are women aged 18-75 years with FIGO 2014 (International Federation of Gynecology and Obstetrics) stage IB2-IIB disease with lymph node positivity or stage III-IVA disease. Patients will be randomly assigned to two groups. Patients in the control group will receive serplulimab immunotherapy combined with concurrent chemoradiotherapy, followed by maintenance serplulimab for up to 2 years. Patients in the experimental group will receive, in addition to the above treatment, two cycles of induction chemotherapy and four cycles of consolidation chemotherapy, consisting of paclitaxel and platinum-based agents. The primary endpoint of this study is progression-free survival (PFS), which will be assessed by investigators according to RECIST version 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily willing to participate in the clinical study, fully informed about the study, and signed the informed consent form (ICF);
2. Willing and able to comply with all study procedures;
3. Female aged 18-75 years;
4. ECOG performance status of 0 or 1;
5. PD-L1 status not restricted;
6. Histologically confirmed cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma;
7. FIGO 2014 (International Federation of Gynecology and Obstetrics) stage IB2-IIB with positive lymph nodes, or stage III-IVA;
8. Patients must meet the following hematologic, renal, and hepatic function criteria:
9. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count ≥ 100 × 10⁹/L; Total bilirubin, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 1.5 × upper limit of normal (ULN); Serum creatinine ≤ upper limit of normal (ULN); No prior anti-tumor treatment; Expected survival > 6 months;
10. Female subjects must have a negative serum pregnancy test within 14 days prior to study treatment, agree to use effective contraception during treatment and for 6 months after treatment, and breastfeeding is prohibited during the study.

Exclusion Criteria:

1. Histologically confirmed small cell cervical cancer;
2. Recurrent cervical cancer or presence of distant metastases;
3. Prior anti-tumor treatment;
4. Current or history of another active, untreated malignancy within the past 5 years, except for adequately treated basal cell carcinoma of the skin or carcinoma in situ;
5. Any active or known autoimmune disease;
6. Active infection;
7. Requirement for systemic treatment with corticosteroids or other immunosuppressive agents within 14 days prior to randomization;
8. Arterial or venous thromboembolic events within 6 months prior to enrollment;
9. Uncontrolled clinically significant cardiac symptoms or disease;
10. Known allergy to the investigational drug or any of its excipients, or prior severe allergic reaction to other monoclonal antibodies;
11. Pregnant or breastfeeding women;
12. Neurological or psychiatric abnormalities affecting cognitive function;
13. Any other condition or situation that, in the investigator's judgment, would pose a serious risk to the subject's safety, potentially confound study results, or interfere with the subject's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 2 year
  defined as the time from randomization to the first occurrence of disease progression or death from any cause.
OS | through study completion, an average of 2 year
  The time from random assignment to death because of any cause.

SECONDARY OUTCOMES:
safety assessment | through study completion, an average of 2 year
  Adverse events occurring throughout the study period will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Maobin Meng, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital,, Tianjin, Tianjin Municipality, China